CLINICAL TRIAL: NCT01378091
Title: Phase I Open-Label, Dose Escalation Study To Determine The Maximum Tolerated Dose And To Evaluate The Safety Profile of Lenalidomide (Revlimid® CC-5013) With Every Three Week Docetaxel (Taxotere®) In Subjects With Androgen Independent Prostate Cancer
Brief Title: Study of Lenalidomide and Docetaxel in Subjects With Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB3212
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Androgen Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, Docetaxel, Prednisone (Experimental): Subjects will receive this drug combination during a treatment phase and an extension phase.
  Interventions: Drug: Lenalidomide; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Lenalidomide — Supplied as 5 mg and 25 mg capsules.
  The lenalidomide dose levels to be studied include 10, 15, 20, 25, 30, 35 and 40 mg/day.
  Other Names: Revlimid
Drug: Docetaxel — Docetaxel is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug.
  Doses of docetaxel to be studied include 60 and 75 mg/m2 once every three weeks.
  Other Names: Taxotere®
Drug: Prednisone — Prednisone is a synthetic corticosteroid drug that is particularly effective as an immunosuppressant drug.
  5 mg BID daily.
  Other Names: Deltasone

SUMMARY:
Primary objectives:

To determine the maximum tolerated doses (MTDs) of daily lenalidomide and docetaxel given every three weeks and prednisone, as combination therapy to subjects with androgen independent prostate cancer

To evaluate the safety profile of the combination of daily lenalidomide and every three week docetaxel and prednisone when given to subjects with androgen independent prostate cancer

Secondary objective:

To explore the anti-tumor activity of the combination of daily lenalidomide and every 3 week docetaxel and prednisone when given to subjects with androgen independent prostate cancer.

DETAILED DESCRIPTION:
Adenocarcinoma of the prostate is the second leading cause of cancer death in men. There is medication available to help treat this disease, which typically lengthens life by 10 to 12 months. More recent studies have shown average survivals of 20 to 23 months.

The investigators hope that the experimental (research) drug called lenalidomide (Revlimid®), which is being used in this study, will lengthen the lives of these patients by even more time. A different drug in the same drug family has demonstrated activity against a variety of solid tumors as well as hematological malignances. It works against cancer in different ways than chemotherapy by affecting the immune system (the body's ability to naturally fight disease).

The investigators believe that the study drug helps build up patients' immune systems than some of the other popular drugs on the market, and may potentially increase survival rates for patients with hormone refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must understand and voluntarily sign an informed consent document.
* Age > 18 years at the time of signing informed consent form.
* Histological documentation of prostate cancer.
* Subjects must be able to adhere to the study visit schedule and other protocol requirements.
* Radiographic or clinical evidence of measurable or evaluable androgen independent prostate cancer stages D1 or D2.
* Patients must be surgically or medically castrated. If the method is medical castration, the patient must have a serum testosterone level of <50 ng/dl/. The patient should maintain treatment with LH RH antagonists or agonists.
* Patients must have metastatic prostate cancer unresponsive or refractory to androgen blockade by one or more of the following criteria:

  * Progression of unidimensionally measurable disease.
  * Progression of non measurable disease
  * Rising PSA (absolute value of PSA > 5 mg/ml).
  * Rising PSA is defined as at least 2 consecutive rises in PSA to be documented over the reference value (measure 1). The first rising PSA (measure 2) must be taken at least 7 days after the reference value. A third confirmatory PSA is required, and it must be obtained at least seven days after the second measure. If the third measure does not confirm the rise in PSA, a fourth PSA measure is required to be taken to confirm the rise over the second measure.
* Patients who were treated with antiandrogens such as flutamide, or other hormonal agents such as estrogens, or ketoconazole must have been stopped for at least 28 days prior to enrollment. In the case of nilandron and bicalutamide, treatment with these agents must have stopped at least 42 days prior to treatment. If the patient is being treated with corticosteroids, the dose should be stable for 14 days prior to study entry
* ECOG performance status of ≤2 (Appendix I: ECOG Performance Status Scale).
* Regarding Lenalidomide: Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix V: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix VI: Education and Counseling Guidance Document.
* Laboratory values as indicated below:

  * Serum Creatinine <2.0 mg/dL
  * Absolute Neutrophil Count ≥1,500/mm3 (or 1.5 X109/L)
  * Platelet Count >100,000/mm3 (or 100 x 109/L)
  * Aspartate Aminotransferase (AST/SGOT) ≤ 1.5 x upper limit of normal (ULN)
  * Alkaline Phosphatase < 2.5 x ULN (In the absence of liver metastasis, elevated alk phos due to bone mets is permitted)
  * Conjugated Bilirubin < ULN

Exclusion Criteria:

* Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent.
* More than 2 prior regimens of chemotherapy.
* Use of thalidomide or biologic response modifier therapy within 28 days of initiation of therapy
* Prior desquamating rash while taking thalidomide therapy.
* Prior > grade-2 allergic reaction to thalidomide.
* Any prior use of lenalidomide. Subjects may have received prior thalidomide therapy.
* Concurrent use of any other anti-cancer agents, excluding bisphosphonates.
* Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
* Active infection, known positive for HIV or hepatitis B or C.
* Known hypersensitivity or intolerance to taxanes or polysorbate 80.
* Known hypersensitivity reaction to thalidomide
* Use of any other experimental drug or therapy within 28 days.
* Subjects with > grade-2 neuropathy.
* Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the breast, or superficial bladder cancer) unless the subject has been free of disease for > 3 years.
* Prior whole pelvic radiation, or prior treatment with strontium. Prior treatment with samarium is permitted.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of lenalidomide | Up to 2 years
  The MTDs of lenalidomide, docetaxel and prednisone when given as combination therapy will be defined as the highest dose level at which no more than 1 out of 6 subjects experiences Dose Limiting Toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Edward Gelmann, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Cornell Weill Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided